CLINICAL TRIAL: NCT00638040
Title: The Gene Expression Studies of Tumor Microenvironments and Their Roles in Tumor Progression
Brief Title: The Gene Expression Studies of the Role of Tumor Microenvironments in Tumor Progression
Status: Withdrawn | Type: Observational
Why Stopped: the study has stopped due to no recruitment
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Other Study IDs: Pro00006979; R01CA125618 (NIH); 9070-07
Record Dates: First submitted 2008-03-12; First posted 2008-03-18 (Estimated); Last update posted 2014-07-11 (Estimated); Status verified 2013-02

CONDITIONS: Hypoxia; Lactic Acidosis
Keywords: hypoxia; lactate; pH; tumor microenvironments; survival
MeSH Terms: conditions — Hypoxia; Acidosis, Lactic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- 1: The purpose of this study is to analyze the gene expression patterns associated with various microenvironmental stresses in tumors to understand their roles in tumor progression and treatment responses. To achieve this goal, we will perform gene expression analysis of the tumor samples collected from an IRB-approved study (IRB #: 4516-05-2R2) International Phase III Study of Chemoradiotherapy versus Chemoradiotherapy Plus Hyperthermia for Locally Advanced Cervical Cancer directed by Dr. Mark Dewhirst. We will correlate the gene expression signatures of different microenvironmental stresses with the measured physiological parameters to understand their role in tumor progression, treatment response and clinical outcomes.

SUMMARY:
The purpose of this study is to analyze the gene expression patterns associated with various microenvironmental stresses in tumors to understand their roles in tumor progression and treatment responses. To achieve this goal, we will perform gene expression analysis of the tumor samples collected from an IRB-approved study (IRB #: 4516-05-2R2) International Phase III Study of Chemoradiotherapy versus Chemoradiotherapy Plus Hyperthermia for Locally Advanced Cervical Cancer directed by Dr. Mark Dewhirst. We will correlate the gene expression signatures of different microenvironmental stresses with the measured physiological parameters to understand their role in tumor progression, treatment response and clinical outcomes.

DETAILED DESCRIPTION:
In the first part of the proposal, we will determine the cellular responses to various microenvironmental factors (such as lactosis, acidosis, hypoxia, glucose deprivation) in cultured epithelial cells (commercially obtained) making use of DNA microarray analysis. From the analysis of these microarray assays, we will obtain the gene signatures reflecting how cells respond to these environments stresses. These gene signatures will be used to analyze and annotate the gene expression patterns in the tumor samples and whether hyperthermia will affect the physiological parameters and the corresponding gene signatures.

In the second part of the proposal, we will work with Dr. Dewhirst to perform gene expression study of cervical cancer samples from a phase III, multicenter, randomized clinical trial (IRB 4516-05-2R2). The subjects will de-identified and we will not obtain directly the PHI of the subjects in this trial. Subjects will be randomized to chemoradiotherapy alone or chemoradiotherapy + hyperthermia. For subjects randomized to hyperthermia, heat treatments will be administered concurrently with chemotherapy once weekly during the course of external beam radiation. In the hyperthermia suite, catheters will be placed in the cervical os, vagina and rectum for internal temperature monitoring. Hyperthermia will be given externally to the pelvis and abdomen using the BSD Sigma 60 ,Sigma Eye or Sigma Ellipse systems. Initial power will be limited to less than 1500 watts with phase and amplitude adjusted for equal surface electric fields in each quadrant of the applicator. Heating will continue for 60 minutes after average cervical os or interstitial temperatures of 40°C have been achieved, or for a maximum total duration of 90 minutes, whichever is longest. The bolus temperature will be 37° at initiation of power and will be reduced as necessary for patient comfort and/or to help maintain oral temperature of 38.5C. Power will also be reduced or treatment will be stopped at the patient request, or due to intractable pain, nausea or vomiting, if normal tissue temperature rises to 44°C, pulse > 160, BP > 180/100 or < 90/50, altered mental status, or systemic temperature > 38.5°C.

A. The research materials will include the tumor biopsy obtained before and after HT treatments to be used for gene expression studies as well as for the IHC and ISH studies to the findings from our microarray analysis. We will also obtain the information on the tumor physiological parameters information measured in these tumors.

B. The data of the tumor physiological parameters measured and the response to treatments and other clinical outcomes of these patients will also be acquired.

C. Only the physicians taking care of the patients will have access to the patient identifies and other Protected Health Information (PHI). All information will be de-identified and remain anonymous during the studies.

D. The specimens will be collected when the patients undergo medical care for their respective diseases. No new materials or data will need to be collected specifically for this proposal. These biopsies and physiological measurements are included in the original proposed clinical trials.

ELIGIBILITY:
Inclusion Criteria:

* Invasive cervical carcinoma (small cell histology excluded)
* Age 18 or over
* FIGO stage IIb-IVa
* ECOG/WHO 0,1, or 2, or >/= 70% respectively
* WBC >/= 3,000, platelets >/= 100,000
* Hgb>12.0 g/dL or >7.5 mmol/L, with transfusion if needed
* Serum bilirubin </= 1.5 times ULN, transaminase </= 3 times ULN
* Calculated creatinine clearance > 60 ml/liter (Cockcroft)
* Para-aortic adenopathy absent or 1.5 cm in greatest dimension on CT/MRI
* No history of myocardial infarction in the last 6 months
* No symptomatic angina pectoris
* Any past history of coronary artery disease must require assessment and clearance by the PCP and/or cardiologist
* Negative pregnancy test in patients under 50
* Written informed consent

Exclusion Criteria:

* Patients who have undergone surgical resection of the primary tumor are not eligible (Limited surgical resection of pelvic nodes without TAH is acceptable)
* Patients with pacemakers or implanted defibrillators
* Patients with significant metallic foreign bodies (i.e. hip replacements, bone metallic rods, orthopedic plates, etc.)
* Prior radiotherapy or chemotherapy

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: The subjects will be de-identified and a system of patient identified will be used to correlate with the clinical data. The patients will be recruited as described in the original approved study. When patients with newly diagnosed cervix cancer are seen at Duke in the GYN Oncology Division or Radiation Oncology, appropriate patients will be offered protocol enrollment. Clinical faculty in both divisions also see new patients at satellite clinics elsewhere in North Carolina and Virginia, and eligible patients may also be enrolled from these encounters. We anticipate enrolling significant number of Spanish speaking women having in mind the increased growth of Latino population in the area.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2009-09; Primary Completion 2012-09 (Actual); Study Completion 2012-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jen-Tsan Chi, Ph.D., Principal Investigator — Duke University
Locations (1):
- Duke Medical Center, Durham, North Carolina, United States